CLINICAL TRIAL: NCT01667042
Title: Scleroderma Lung: Role of Gastroesophageal Reflux, Microaspiration and Cough
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Augustine S. Lee, M.D., Mayo Clinic
Other Study IDs: 12-000304
Record Dates: First submitted 2012-08-14; First posted 2012-08-17 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Scleroderma Lung
Keywords: Scleroderma Lung; Gastroesophageal Reflux; Microaspiration; Cough
MeSH Terms: conditions — Gastroesophageal Reflux; Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Without Interstitial lung disease (ILD)
- With Interstitial lung disease (ILD)

SUMMARY:
This is a mechanistic research study to evaluate the relationship between cough, reflux, and aspiration in patients with systemic sclerosis (scleroderma).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years old.
* Fulfilling the American College of Rheumatology criteria for SSc.
* For ILD subgroup (n=6):

  * An upright chest-roentgenogram (chest x-ray) is abnormal and compatible with an interstitial lung disease.
  * HRCT of the chest confirms the presence of bilateral reticular, ground glass, and/or honeycomb abnormalities that is otherwise unexplained by an alternative process
  * The HRCT fibrosis score must be ≥ 7.
  * The total lung capacity (TLC, measured by body plethysmography) and/or the diffusing capacity of the lung for carbon monoxide (DLCO) is below the predicted normal.
  * The forced vital capacity (FVC) is reduced below the predicted normal.
  * The patient is symptomatic (i.e. dyspnea and/or a chronic cough) for more than 8 weeks that is otherwise unexplained by an alternative mechanism.
* For No ILD subgroup (n=6):

  * No radiographic evidence of ILD on plain chest x-ray.
  * The HRCT fibrosis score, when performed) must be < 7
  * The TLC and FVC are within their predicted normal.
  * The DLCO is within the predicted normal, except when reduced in isolation by pulmonary hypertension.

Exclusion Criteria:

* Active smoking within the 6 months.
* Pneumonia or bronchitis in past 4 weeks.
* Active acute illness such as uncontrolled heart failure, infection, or asthma.
* Use of more than 3 liters per minute (LPM) of oxygen by nasal cannula at rest.
* Coordinator, investigator, or clinician concerns on the patient's compliance, safety, or in ability to complete study requirements.
* Morbid condition not expected to live more than 1 year.
* Alternative cause or diagnosis for the patient's ILD besides SSc.
* Pregnancy.
* Obstructive lung disease with an FEV1 (forced expiratory volume in 1 second) to FVC ratio less than 0.7, nor radiographic evidence of emphysema on CT.
* Planned therapeutic procedures involving the esophagus (e.g. dilation, surgery) prior to completion of study tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive adult patients seen at the Mayo Clinic in Florida with a confirmed diagnosis of systemic sclerosis (SSc) will be eligible.
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2012-08; Primary Completion 2014-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Airway pepsin concentration | cross-sectional
  Cross-sectional comparison between airway pepsin level, cough frequency, FVC, DLCO, and CT fibrosis score

CONTACTS AND LOCATIONS:
Overall Officials: Augustine Lee, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States